CLINICAL TRIAL: NCT06234787
Title: Continuous Subcutaneous Glucose Monitoring: A Descriptive Study of Its Use in Critical Patients
Brief Title: Continuous Subcutaneous Glucose Monitoring in Critical Patients
Status: Recruiting | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Samuel Gonzalez Lopez, Principal Investigator, Universidad Europea de Madrid
Other Study IDs: MCGUCI1
Record Dates: First submitted 2023-12-17; First posted 2024-01-31 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Hyperglycemia; Hypoglycemia; Diabetes; Critical Care; Critically Ill Patients
Keywords: continuous subcutaneous glucose monitoring; critical care; intensive care; hypoglycemia
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patients: Patients admitted to the Intensive Care Unit (ICU) at HLA Moncloa Hospital

SUMMARY:
This is a single-center, observational, descriptive, longitudinal, and prospective study This study aims to determine the cumulative incidence during admission and the incidence rate of potential hypoglycemic events (defined as subcutaneous glucose <80 mg/dL detected by CGM) in patients admitted to the Intensive Care Unit (ICU) of HLA Moncloa Hospital over four years of follow-up. The study also aims to document the occurrences of hypoglycemic events, describe the characteristics of patients receiving CGM sensors, and outline the actions taken as a result of detecting potential hypoglycemic events

DETAILED DESCRIPTION:
The disturbances in glycemic control, including type 1 and type 2 diabetes, are increasingly prevalent in the general population, with estimates suggesting that this trend will continue for at least the next 20 years. Critically ill patients are particularly predisposed to glycemic alterations due, among other factors, to stress, fasting, infections, and administered treatments.

Hyperglycemia is detrimental to critically ill patients. Sustainedly elevated blood glucose levels lead to immunosuppression, hindering leukocyte function, reducing phagocytic capacity, and altering complement function. Furthermore, hyperglycemia enhances proinflammatory mechanisms and oxidative stress. Hemodynamic management is also affected, resulting in endothelial dysfunction and osmotic diuresis, promoting dehydration, electrolyte imbalances, and tissue hypoperfusion.

For this reason, most current recommendations for glycemic control in critically ill patients advise insulin treatment when blood glucose levels exceed 180 mg/dL. However, the ideal glucose range for maintaining patients is still a subject of debate because, despite knowing that hyperglycemia is harmful, its treatment carries a high risk of hypoglycemia. Severe hypoglycemia (glucose <40 mg/dL) increases the risk of death by more than three times in critically ill patients.

The incidence of hypoglycemia in critically ill patients varies widely depending on the type of patient and the protocol used for hyperglycemia control. Generally, it is estimated that between 3% and 20% of critically ill patients may experience severe hypoglycemia during their hospitalization. On the other hand, hypoglycemia can be easily prevented or treated in hospitalized patients through the infusion of glucose solutions if identified correctly.

In recent years, the use of continuous subcutaneous glucose monitoring (CGM) sensors has revolutionized clinical practice for non-hospitalized diabetic patients. Subcutaneous glucose is directly related to capillary blood glucose and arterial blood glucose, so changes in blood glucose concentration will be transmitted to subcutaneous tissue within the next 5 to 10 minutes. CGM in critically ill patients has been shown to significantly reduce the incidence of hypoglycemia, mortality, and glycemic variability compared to standard practice.

Given the current evidence, the Intensive Care Unit (ICU) at HLA Moncloa University Hospital has developed a guide for the use of CGM sensors in critically ill patients receiving insulin treatment, with the primary goal of reducing episodes of severe hypoglycemia in these patients. This guide has been in use since May 2023 (see ANNEX).

The main utility of these sensors in critically ill patients is to detect individuals at risk of experiencing hypoglycemia, which the investigators may consider potential hypoglycemic events. However, to the best of our knowledge, there is currently no unified clinical practice regarding the use of these devices in critically ill patients, and it is not possible to find clinical practice guidelines or recommendations for the detection thresholds of potential hypoglycemic events or studies describing the characteristics of these events.

Design:

This is a single-center, observational, descriptive, longitudinal, and prospective study.

Scope and Study Population:

The study will be conducted on patients admitted to the ICU at HLA Moncloa Hospital over the course of four years.

Procedures:

All patients admitted to the Intensive Care Unit (ICU) who are potential candidates for inclusion in the study will be informed about it, and their informed consent will be requested.

If patients agree to participate, the inclusion criteria will be ensured. Therefore, a continuous glucose monitoring sensor will be placed according to the detailed instructions in Annex 1.

Patients will receive treatments according to the center's usual clinical practice and following the criteria of their responsible physician based on the patient's characteristics in each case.

The device records glucose readings every 5 minutes. The information is automatically recorded on the reading device.

If at any time the device detects a potential hypoglycemia, healthcare personnel will act according to the device placement guide (ANNEX 1), which details the procedure to follow. If confirmed, corrections will be made according to the criteria of the responsible physician.

At the time of patient discharge or death, the principal investigator will review the patient medical history to create a pseudonymized database that includes the patient study variables, treatments, and duration of ICU stay, as well as the glucose records made by the continuous monitoring device. This information will be stored for 5 years on the hospital intranet server, along with other confidential information from the ICU at HLA Moncloa Hospital.

Alarms:

Alarms will be set up with the Freestyle Libre 2 sensor reader similarly for all patients.

Low glucose alarm (subcutaneous glucose <80 mg/dL):

After the alarm, capillary, arterial, or venous blood glucose will be checked, and actions will be taken according to the standard protocol of the ICU at HLA Moncloa Hospital.

Definitions of hypoglycemia:

Potential Hypoglycemia: Any continuous subcutaneous glucose measurement below 80 mg/dL confirmed by checking capillary, arterial, or venous blood glucose values up to 90 mg/dL (a margin of 10 mg/dL difference between subcutaneous glucose and blood glucose obtained will be accepted for hypoglycemia confirmation).

Severe Hypoglycemia: Any glucose measurement below 40 mg/dL, whether in capillary, arterial, or venous blood.

Moderate Hypoglycemia: Any glucose measurement between 40 and 54 mg/dL, whether in capillary, arterial, or venous blood.

Mild Hypoglycemia: Any glucose measurement between 55 and 69 mg/dL, whether in capillary, arterial, or venous blood.

False Hypoglycemia: Any continuous subcutaneous glucose measurement below 80 mg/dL is discarded by checking capillary, arterial, or venous blood glucose values above 90 mg/dL.

Capillary, Arterial, and Venous Glucose:

Critically ill patients routinely undergo glucose determinations several times throughout the day and in response to specific symptoms (dizziness, fatigue, weakness, headaches, confusion, speech disturbances, blurred vision, seizures, and coma). This includes capillary glucose measurements at the bedside, arterial blood gas analyses, or laboratory blood glucose tests on arterial or venous blood.

The results of all glucose determinations performed on the patient will be systematically recorded. This way, the incidence and incidence rate of mild, moderate, and severe hypoglycemia occurring during hospitalization will be documented.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in patients admitted to the ICU of HLA Moncloa Hospital over four years. Patients admitted to the ICU, undergoing insulin treatment, and having a CGM sensor.
* Patients who sign the voluntary consent to participate in the study (Annex 2). If the participant is not in full physical or intellectual capacity to provide their signature on the informed consent, the responsible investigator will request such consent from their direct family member or the person legally designated to make decisions on their behalf regarding health matters. This measure is taken to ensure that the participant's rights are respected, and the integrity of the consent process is maintained, even in situations where their decision-making capacity may be compromised.

Exclusion Criteria:

* Patients from whom information on CGM cannot be obtained for technical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU, undergoing insulin treatment, and having a CGM sensor
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the cumulative incidence or risk of potential hypoglycemia during ICU admission | 4 years
  To determine the cumulative incidence or risk of potential hypoglycemia during ICU admission (cases of potential hypoglycemia/number of patients x 100) and the incidence rate (cases of potential hypoglycemia/1000 x patient x hour) in critically ill patients undergoing insulin treatment using CGM sensors. The investigators will consider potential hypoglycemia any instance where the CGM sensor indicates low glucose (glucose <80 mg/dL)

SECONDARY OUTCOMES:
To determine the incidence of severe hypoglycemia | 4 years
  To determine the incidence of severe hypoglycemia (glucose <40 mg/dL), moderate (glucose between 40 and 55 mg/dL), or mild (glucose between 56 and 70 mg/dL) (cases of hypoglycemia/number of patients x 100) during the ICU stay and the incidence rates (cases of hypoglycemia/1000 patients x hour) in critically ill patients undergoing insulin treatment using CGM sensors.
To determine the percentage of false potential hypoglycemia | 4 years
  To determine the percentage of false potential hypoglycemia, understood as warnings for potential hypoglycemia that do not correspond to low capillary glucose values (glucose <90 mg/dL)
To describe the type of patients admitted to the ICU who are equipped with a CGM sensor | 4 years
  To describe the type of patients admitted to the ICU who are equipped with a CGM sensor in our unit.
To describe the glycemic profile of critically ill patients | 4 years
  To describe the glycemic profile of critically ill patients undergoing insulin treatment (Maximum glucose, minimum glucose, average glucose, glycemic variability, time in range, Hb A1c, diet used, insulin requirement, insulin protocol employed).
To describe the actions taken by healthcare personnel after a potential hypoglycemia alarm | 4 years
  To describe the actions taken by healthcare personnel after a potential hypoglycemia alarm (administration of intravenous glucose (iv) glucosmon 50% in ml, administration of iv glucose glucosmon 33% in ml, initiation of iv glucose infusion 5% ml/h, iv glucose infusion 10% (ml/h), others).
To describe the theoretical cumulative incidence of potential hypoglycemia with alternative thresholds of 70, 75, 85, or 90 mg/dL | 4 years
  To describe the theoretical cumulative incidence of potential hypoglycemia with alternative thresholds of 70, 75, 85, or 90 mg/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario HLA Moncloa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT06234787/Prot_002.pdf
  • Informed Consent Form (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT06234787/ICF_001.pdf